CLINICAL TRIAL: NCT05169632
Title: Combined Cognitive and Physical Training for the Neurorehabilitation of Executive Deficits After Stroke: an Exploratory Randomized Controlled Trial
Brief Title: Computerized Cognitive Rehabilitation of Executive Deficits in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Prof. Arseny Sokolov, MD, PhD, Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHUV-DNC-CCT-STROKE-2021
Record Dates: First submitted 2021-10-29; First posted 2021-12-27 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Executive Dysfunction
Keywords: Stroke Rehabilitation; Neurological Rehabilitation; Exercise Therapy; Brain Training; Nervous System Diseases; Neurocognitive Disorders; Cognition Disorders; Mental Disorders; Vascular System Injuries; Cerebrovascular Disorders; Multimodal Intervention; e-Health; Digital Intervention; Exergame
MeSH Terms: conditions — Stroke; Nervous System Diseases; Neurocognitive Disorders; Cognition Disorders; Mental Disorders; Vascular System Injuries; Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (CTR) (Active Comparator): Computerized Gaming Rehabilitation Program 1
  Interventions: Device: Computerized Gaming Rehabilitation Program 1
- Intervention group (INT) (Experimental): Computerized Gaming Rehabilitation Program 2
  Interventions: Device: Computerized Gaming Rehabilitation Program 2

INTERVENTIONS:
Device: Computerized Gaming Rehabilitation Program 1 — Brain training games with physical exercise component.
  Arms: Control group (CTR)
Device: Computerized Gaming Rehabilitation Program 2 — Cognitive training games with physical exercise component.
  Arms: Intervention group (INT)

SUMMARY:
WHO: 32 participants with executive deficits related to a stroke, able to engage in moderate physical activity.

WHY: Around one third of stroke patients suffer from cognitive deficits in the long term, which have a detrimental impact on everyday personal and professional life. The purpose of this study is to evaluate two sets of computerized exercises combining cognitive and physical effort to see if they can improve executive function.

WHAT: Study participants first undergo cognitive and physical assessments. Additional questionnaires will assess mood, everyday life cognition, function and quality. This will be followed by a 6 week training period with 3 training sessions a week. The effect of the cognitive and physical training will be measured in a post-training evaluation session. Six months after completion of the training, the study will evaluate cognitive and physical abilities of participants to study long-term effects of the respective training program.

WHERE: Both the evaluation and the training sessions will be conducted on the premises of the Centre Hospitalier Universitaire Vaudoise (Pavillon 4, Avenue de Beaumont, 1005 Lausanne, Switzerland)

DETAILED DESCRIPTION:
This is an exploratory Randomized Controlled Trial with the purpose of evaluating the potential of two sets of gamified cognitive and physical exercises in the neurorehabilitation of cognitive deficits following a stroke.

Upon recruitment, eligible study participants (see 'Eligibility Criteria') receive a detailed oral and written description about the scientific background, aims and methods of the study. Additional information will be provided about potential benefits and risks associated with study participation, as well as about the voluntary nature of participation throughout the study. The participant's written informed consent is required for study enrollment.

After inclusion in the study, participants are randomized into one of two different training programs with equal chance of attribution and without possibility of choosing:

* Program 1 involves brain training games with a physical exercise component.
* Program 2 involves cognitive training games with a physical exercise component.

Independently of program attribution, participants engage in a pre-training assessment, a six-week training period, a post-training assessment and a 6-month-follow-up assessment. The three assessments include on-site cognitive and physical evaluation, along with the completion of self-report questionnaires concerning subjective cognitive function, mood, and quality of life.

Following the first assessment, study participants engage in a 6-week training period. In both programs, participants engage in 3 weekly trainings of 90 minutes duration each.

A final follow-up visit is scheduled 6 months after the completion of the last training session. The cognitive and physical testing together with the questionnaires will be repeated to examine the long-term effects of the training programs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ischemic or haemorrhagic cerebral stroke ≥ 8 weeks before study inclusion
* Cognitive complaint and/or clinical impression of dysexecutive syndrome
* Z-Score < -1.0 in at least two of the following domains

  * Cognitive flexibility (Trail-Making Test B/A)
  * Cognitive interference (Stroop color word interference task)
  * Divided attention (TAP divided attention)
  * Working memory (TAP working memory, Forward Digit Span, Backward Digit Span)
  * Design fluency (Five-points test)

Exclusion Criteria:

* Major neurocognitive disorder according to the DSM-5
* Proximal extremity paresis grade < M4 on the Medical Research Council (MRC) Scale for Muscle Strength in at least one of four extremities
* Insufficient visual acuity, visual field or hemispatial attention to engage in the training
* Inability to discriminate colour: < 12 points on the Ishihara test
* Changes over the last 4 weeks in antidepressive, anxiolytic or in acetylcholinesterase inhibitor drugs
* Thoracic pain and/or heart palpitations at rest, during or following a physical effort (based on self-report)
* Clinically unstable cardio-vascular disease
* Falls in the past 12 weeks as evaluated in the enrolment interview [Hopkins Falls Grading Scale (Grade >1)]
* High risk of falling according to a score of over 15 seconds on the Four Square Step Test (FSST)
* Insufficient knowledge or capacity of French to follow instructions
* Incapacity or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive interference after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Cognitive interference is measured using the Delis-Kaplan Executive Function System (D-KEFS; Delis, Kaplan, Kramer, 2001) Stroop Test
Change in divided attention after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Divided attention is measured using the Test of Attentional Performance (TAP, version 2.3.1; Zimmermann and Fimm, 2002) subtest for divided attention
Change in visuospatial short term memory after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Visuospatial short term memory is measured by the immediate recall of the Brief Visuospatial Memory Test-Revised (BVMT-R; Benedict, 1996)
Change in subjective executive function after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Subjective executive function is measured by the Working Memory Questionnaire (WMQ; Vallat-Azouvi et al, 2012; 30 items, participants rate 10 statements on storage, attention and executive domain on a Likert-scale from 1-5 (not at all - extremely))

SECONDARY OUTCOMES:
Change in visual working memory after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Visual working memory will be assessed via performance on the computerized 'Filter task' (Vogel, 2005).
Change in design fluency after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  The Five-Point Test (Regard, 1982) will be used to assess design fluency.
Change in processing speed after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  The Trail-Making-Test Part A (Reitan, 1955) will be used to assess processing speed.
Change in cognitive flexibility assessed by the TMT-B after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Cognitive flexibility will be measured using the Trail-Making-Test B (TMT-B; Reitan, 1955).
Change in cognitive flexibility assessed by the TAP Flexibility after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Cognitive flexibility will be measured using the subscale 'Flexibility' of the Test of Attentional Performance (TAP, version 2.3.1; Zimmermann and Fimm, 2002)
Change in cognitive inhibition after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  The Test of Attentional Performance (TAP, version 2.3.1; Zimmermann and Fimm, 2002) subtest Go/NoGo will assess cognitive inhibition.
Change in cognitive multitasking after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  A subtest of a custom-made tablet-based cognitive evaluation tool will measure cognitive multitasking.
Change in covert shift of attention after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Measured by the corresponding subtest of the Test of Attentional Performance (TAP, version 2.3.1; Zimmermann and Fimm, 2002).
Change in risk of falls and postural stability after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Postural stability and risk of falls will be assessed using the BTrackS Balance Plate (FDA registered class 1 medical device #3010668481)
Change in dynamic stability after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Dynamic stability will be assessed by the Four Square Step Test (FSST; Dite et al, 2002), which tests the participant's ability to step over objects forwards, sideways and backwards; the movements of the FSST are comparable to the ones implemented in the training program.
Change in ability to perform a cognitive and physical dual task after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  In order to assess cognitive and motor dual task ability, the study participant will perform the 'Timed Up and Go Cognitive' subtest from the MiniBESTest (Franchignoni et al, 2010).
Change in heart rate after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Heart rate (HR) will be recorded at rest in supine position during a 5-minute window using a chest belt.
Change in heart rate variability after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Heart rate variability (HRv) will be recorded at rest in supine position during a 5-minute window using a chest belt.
Change in systolic and diastolic blood pressure after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Determined by the mean of three blood pressure measurements using a sphygmomanometer and a stethoscope.
Everyday physical activity during 6-week training period. | 6 weeks
  Measuring daily step count and minutes of daily activity using a wrist-attached wearable device will determine everyday physical acitivity during the training period.
Change in everyday life quality after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Study participants will rate everyday life quality using the Quality of Life after Brain Injury questionnaire (QOLIBRI; von Steinbuchel, 2010; 36 items originally, adapted to 35 items for stroke, participants rate applicability of statements on quality of life after stroke from not at all to very))
Change in everyday life cognitive function after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Study participants will rate everyday life cognitive function using the Cognitive Failure Questionnaire (CFQ; Broadbent, 1982; 25 items, participants rate the frequency of situations representing cognitive dysfunction in the past 6 months from very often (4 points) to never (0 points), a lower score represents a better subjective cognitive function).
Change in mood after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Mood is measured by the Hospital Anxiety and Depression Scale (HAD-S; Zigmond and Snaith, 1983), which tests for both anxiety and depression in a 14-item questionnaire (7 items each, participants rate statements on a Likert-Scale from 0-3 for each statement, the maximal score is 28 for each domain, the cut-off 11 for anxiety and depression is points or more).
Change in apathy after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Study participants will rate their degree of apathy using the self-administered Dimensional Apathy Scale (DAS; 24 items; Radakovic and Abrahams, 2014).
Change in fatigue after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Study participants will rate their degree of fatigue on the Modified Fatigue Impact Scale (MFIS; Larson, 2013; 21 items in total, whereof 9 items on a physical subscale, 10 items on a cognitive subscale and 2 items on a psychosocial subscale; every item contains a statement rated on a Likert-Scale from 0-4 (never - almost always), a higher score represents a greater impact of fatigue on the participant's life)
Change in subjective balance after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  The subjective balance of study participants will be measured using the Tinetti Falls Efficacy scale (Tinetti, 1990), a 10-item questionnaire.

OTHER OUTCOMES:
Subjective experience with technology used in study | 6 weeks
  Regardless of training group attribution, study participants will rate the user-friendliness and the experience of the training using the 10-item System Usability Scale (Brooke, 1996; 10 statements about system usability rated on a Likert-scale from 1-5 (strongly disagree - strongly agree)).
Perception of game training | 6 weeks
  Regardless of training group attribution, study participants will rate their perception of game training using the Perception of game training questionnaire (Boot et al, 2013; 4 statements on enjoyment, challenge, frustration and motivation associated with the game, participants rate their agreement with the statement on a Likert-scale from 1 (lowest) to 7 (highest)).

CONTACTS AND LOCATIONS:
Overall Officials: Arseny A. Sokolov, Prof MD PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland; Giulia Binarelli, PhD, Study Chair — Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland
Locations (1):
- Lausanne University Hospital (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zimmermann, P. and B. Fimm, A test battery for attentional performance. Applied Neuropsychology of Attention, Theory, Diagnosis and Rehabilitation 2002: p. 110-151.
- [Background] Benedict, R.H.B., et al., Revision of the Brief Visuospatial Memory Test: Studies of normal performance, reliability, and Validity. Psychological Assessment, 1996.
- [Background] Delis DC, Kramer JH, Kaplan E, Holdnack J. Reliability and validity of the Delis-Kaplan Executive Function System: an update. J Int Neuropsychol Soc. 2004 Mar;10(2):301-3. doi: 10.1017/S1355617704102191. No abstract available. PMID 15012851
- [Background] Vallat-Azouvi C, Pradat-Diehl P, Azouvi P. The Working Memory Questionnaire: a scale to assess everyday life problems related to deficits of working memory in brain injured patients. Neuropsychol Rehabil. 2012;22(4):634-49. doi: 10.1080/09602011.2012.681110. Epub 2012 Apr 27. PMID 22537095
- [Background] Vogel EK, McCollough AW, Machizawa MG. Neural measures reveal individual differences in controlling access to working memory. Nature. 2005 Nov 24;438(7067):500-3. doi: 10.1038/nature04171. PMID 16306992
- [Background] Regard M, Strauss E, Knapp P. Children's production on verbal and non-verbal fluency tasks. Percept Mot Skills. 1982 Dec;55(3 Pt 1):839-44. doi: 10.2466/pms.1982.55.3.839. No abstract available. PMID 7162920
- [Background] REITAN RM. The relation of the trail making test to organic brain damage. J Consult Psychol. 1955 Oct;19(5):393-4. doi: 10.1037/h0044509. No abstract available. PMID 13263471
- [Background] Dite W, Temple VA. A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil. 2002 Nov;83(11):1566-71. doi: 10.1053/apmr.2002.35469. PMID 12422327
- [Background] Franchignoni F, Horak F, Godi M, Nardone A, Giordano A. Using psychometric techniques to improve the Balance Evaluation Systems Test: the mini-BESTest. J Rehabil Med. 2010 Apr;42(4):323-31. doi: 10.2340/16501977-0537. PMID 20461334
- [Background] von Steinbuchel N, Wilson L, Gibbons H, Hawthorne G, Hofer S, Schmidt S, Bullinger M, Maas A, Neugebauer E, Powell J, von Wild K, Zitnay G, Bakx W, Christensen AL, Koskinen S, Formisano R, Saarajuri J, Sasse N, Truelle JL; QOLIBRI Task Force. Quality of Life after Brain Injury (QOLIBRI): scale validity and correlates of quality of life. J Neurotrauma. 2010 Jul;27(7):1157-65. doi: 10.1089/neu.2009.1077. PMID 20210602
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Radakovic R, Abrahams S. Developing a new apathy measurement scale: Dimensional Apathy Scale. Psychiatry Res. 2014 Nov 30;219(3):658-63. doi: 10.1016/j.psychres.2014.06.010. Epub 2014 Jun 19. PMID 24972546
- [Background] Larson RD. Psychometric properties of the modified fatigue impact scale. Int J MS Care. 2013 Spring;15(1):15-20. doi: 10.7224/1537-2073.2012-019. PMID 24453758
- [Background] Tinetti ME, Richman D, Powell L. Falls efficacy as a measure of fear of falling. J Gerontol. 1990 Nov;45(6):P239-43. doi: 10.1093/geronj/45.6.p239. PMID 2229948
- [Background] Brooke, J., SUS: A 'Quick and Dirty' Usability Scale. 1996.
- [Background] Boot WR, Champion M, Blakely DP, Wright T, Souders DJ, Charness N. Video games as a means to reduce age-related cognitive decline: attitudes, compliance, and effectiveness. Front Psychol. 2013 Feb 1;4:31. doi: 10.3389/fpsyg.2013.00031. eCollection 2013. PMID 23378841